CLINICAL TRIAL: NCT01599156
Title: Reflexology for Patients Suffering From Chronic Constipation- a Phase II B, Single Armed, Open Label Study.
Brief Title: Reflexology for Chronic Constipation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REF11
Record Dates: First submitted 2012-05-06; First posted 2012-05-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Constipation
Keywords: Chronic constipation; Reflexology; Complementary medicine
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reflexology (Experimental): reflexology treatment, x2-3/week for 12 weeks
  Interventions: Procedure: Reflexology

INTERVENTIONS:
Procedure: Reflexology — Reflexology is a therapy whereby diagnosis and treatment are done on the patient's feet. According to reflexology, our feet are a micro-cosmos of our bodies and contain all the body's systems and internal organs. The treatment is palpation and massage of specific reflex points that respond to the body organs. This massage or palpitation of reflex points improves the physical function of the corresponding organ or system

SUMMARY:
The purpose of this study is to examine if the use of reflexology can alleviate chronic constipation. The trial will last 26 week per patient, 2 week of screening period, 12 weeks of treatment and 12 weeks of follow up. Included in the study will be 40 men and women, 18 years of age or older, which are able to comply with the study guidelines; Fewer than three spontaneous bowel movement per week; and one or more of the following symptoms/signs during more than 25% of bowel movements for at least 12 weeks within the preceding 12 months: (1) straining, lumpy or (2) hard stools, and (3) a sensation of incomplete evacuation. Exclusion criteria are: Loose or watery stool in the absence of laxative use for more than 25% of bowel movements during the 12 weeks preceding the trials; Mushy stool defined as a score of 6 on the Bristol Stool Form Scale for any SBM during the baseline period; Rome III criteria for the irritable bowel syndrome; History of pelvic-floor dysfunction; Neurological pathologies; Psychiatric conditions; Chronic use of medication with a gastro intestinal-activity.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-55 years
* Fewer than three SBMs per week (occurring without the use of a laxative, enema, or suppository within the preceding 24 hours)
* One or more of the following symptoms/signs during more than 25% of bowel movements for at least 12 weeks within the preceding 12 months:(1)straining, lumpy or (2) hard stools, and (3)a sensation of incomplete evacuation Six or fewer SBMs/week and fewer than three complete CSBMs/week during the 14-day baseline period.
* Ability to comply with the study guidelines

Exclusion Criteria:

* Loose or watery stool in the absence of laxative use for more than 25% of bowel movements during the 12 weeks preceding the trials.
* Mushy stool defined as a score of 6 on the Bristol Stool Form Scale for any SBM during the baseline period.
* Rome III criteria for the irritable bowel syndrome.
* History of pelvic-floor dysfunction.
* Neurological pathologies
* Psychiatric conditions
* Chronic use of medication with a GI-activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Change in complete spontaneous bowel movements (CSBM)/week from baseline to 24 weeks | 24 weeks
  Will be assessed daily during the 24 weeks of the study
Increase of at least one CSBM per week from baseline for 9 or more weeks during the 24-week treatment period | 24 weeks
  Will be assessed weekly during the 24 weeks of the study

SECONDARY OUTCOMES:
Stool frequency/Week (CSBMs and spontaneous bowel movements (SBMs) | 24 weeks
  Will be assessed weekly during the 24 weeks of the study
Stool consistency/week using the 7- point Bristol Stool Form Scale, during the 24 weeks of the study period | 24 weeks
  Will be assessed weekly during the 24 weeks of the study
Severity of straining using a 5-point ordinal scale (1 indicates not at all; 5 an extreme amount). | 24 weeks
  Will be assessed daily during the 24 weeks of the study
Abdominal discomfort, using a 5-point ordinal scale (1 indicates not at all; 5 an extreme amount) | 24 weeks
  Will be assessed daily during the 24 weeks of the study
Severity of bloating, using a 5-point ordinal scale (1 indicates not at all; 5 an extreme amount) | 24 weeks
  Will be assessed daily during the 24 weeks of the study
Constipation severity (using a 5-point ordinal scale, with higher scores indicating greater severity) | 24 weeks
  Will be assessed weekly during the 24 weeks of the study
Constipation relief (based on a 7-point balanced scale, with 1 indicating complete relief, 4 indicating no change, and 7 indicating very severe constipation) | 24 weeks
  Will be assessed weekly during the 24 weeks of the study
Satisfaction with the trial results, using a 5-point ordinal scale | 24 weeks
  will be assessed at the 12-week visit and at the 24-week visit (at the study end)
Health related quality of life (using the validated Patient Assessment of Constipation Quality of Life instrument (PAC-QOL) | 24 weeks
  will be assessed at baseline; at the 12-week visit and at the 24-week visit (at the study end)
Treatment side effects | 24 weeks
  Will be assessed at baseline, week 12 and week 24 (trial end)

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Oberbaum, MD, Principal Investigator — Menachem Oberbaum, MD, Phone:+972-2-6666395, Email: oberbaum@szmc.org.il; Joseph Lysy, Principal Investigator — Joseph Lysy,Phone: +972-2-6666116 Email: lysyj@szmc.org.il
Locations (1):
- The Center for Integrative Complementary Medicine, Shaare Zedek Medical Center, Jerusalem, Israel